CLINICAL TRIAL: NCT03643874
Title: Cumulative Dose, 2-Way Crossover Study of the Safety and Efficacy of Albuterol Administered by the Halix™ Dry Powder Inhaler Compared With MDI in Subjects With Asthma
Brief Title: Safety and Efficacy of Albuterol Administered by the Halix™ Dry Powder Inhaler in Subjects With Asthma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Concentrx Pharmaceuticals, Inc. (Industry)
Collaborators: PharPoint Research, Inc. (Industry); Kramer Consulting, LLC (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CONX-201
Record Dates: First submitted 2018-08-07; First posted 2018-08-23 (Actual); Last update posted 2019-01-30 (Actual); Status verified 2019-01

CONDITIONS: Asthma
Keywords: Single-dose disposable dry powder inhaler
MeSH Terms: conditions — Asthma | interventions — Albuterol

STUDY DESIGN:
Intervention Model Description: 2-way cumulative dose crossover
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Halix albuterol 90 mcg (Experimental): Cumulative doses of albuterol administered by the Halix albuterol 90 mcg UDDI will given at intervals as: 1 inhalation, then 1 inhalation 30 min later, then 2 inhalations 30 min later, and then 4 inhalations 30 min later.
  Interventions: Drug: Halix albuterol 90 mcg
- Albuterol HFA MDI 90 mcg (Active Comparator): Cumulative doses of albuterol administered by the albuterol HFA albuterol 90 mcg MDI will given at intervals as: 2 inhalations, then 2 inhalations 30 min later, then 4 inhalations 30 min later, and then 8 inhalations 30 min later.
  Interventions: Drug: albuterol HFA MDI 90 mcg

INTERVENTIONS:
Drug: Halix albuterol 90 mcg — albuterol unit dose disposable DPI delivers 90 mcg of albuterol in the excipient lactose with each inhalation. Albuterol 90 mcg will be given on one of the treatment days in cumulative doses up to a total dose of 720 mcg
  Other Names: Halix
  Arms: Halix albuterol 90 mcg
Drug: albuterol HFA MDI 90 mcg — albuterol HFA MDI delivers 90 mcg of albuterol with each inhalation. Albuterol 90 mcg will be given on one of the treatment days in cumulative doses up to a total dose of 1440 mcg
  Other Names: Ventolin
  Arms: Albuterol HFA MDI 90 mcg

SUMMARY:
Male and female subjects with mild to moderate asthma will be recruited to enroll in a 2-way crossover during which escalating doses of albuterol will be administered at 30 minute intervals on a single treatment day. Albuterol will be administered by the Halix albuterol unit dose disposable inhaler on one day and by Ventolin albuterol HFA MDI on the other day. Assignment to device for albuterol delivery will be by random allocation.

DETAILED DESCRIPTION:
Study Design: This is a phase 2A, open label, cumulative dose, randomized 2-way crossover study designed to assess the safety, efficacy, pharmacodynamics, pharmacokinetics (PK), and extrapulmonary pharmacodynamics of cumulative doses of Halix™ albuterol 90mcg compared with cumulative doses of Ventolin HFA MDI. After completing all screening assessments and meeting all eligibility criteria [including SABA-free screening forced expiratory volume in 1 second (FEV1) ≥50% to <85% of that predicted for age, gender, height, and ethnicity], enrolled subjects will withdraw from use of Ventolin MDI with substitution of Atrovent HFA as the only inhaled bronchodilator for at least 72 hours before each of 2 Treatment Days. On each Treatment Day study treatments will consist of single doses of study drug (albuterol) administered at 30-minute intervals as follows:

Halix™ albuterol UDDI - 1 + 1 + 2 + 4 inhalations [90 mcg per inhalation] Ventolin albuterol MDI -- 2 + 2 + 4 + 8 inhalations [90 mcg (1 puff) per inhalation]

The order in which each treatment will be administered to a subject will be based on randomization to one of 2 possible sequences. Equal numbers of subjects will be assigned to each sequence. The beginning of each Treatment Day will be separated by a washout period of at least 72 hours after the preceding Treatment Day; the washout period not to exceed 240 hours. After Treatment Day 2, subjects will be assessed at an End-of-Study (EOS) Visit which will occur 1 to 5 days after the last administration of study drug.

Prior to each Treatment Day, the subject must not have used >8 actuations of (non-study drug) rescue Ventolin MDI on each of 3 or more days during the previous 7 days and must not have used any non-study drug rescue Ventolin MDI during the 72 hours prior to the start of the Treatment Day. The Treatment Day will not proceed if either of these instances has occurred.

Within the 75 minutes prior to the first study drug dose on each of the 2 Treatment Days, the following procedures will be performed: vital signs (BP and HR), ECG, collection of urine for pregnancy test if subject is a WOCBP, collection of blood for baseline glucose, potassium, and PK, and spirometry at 60 minutes and at 30 minutes prior to the anticipated time of first study drug dose. The average of the FEV1 at 60 minutes and 30 minutes prior to the first study drug dose on Treatment Day 1 must be ≥ 50% and < 85% of percent predicted in order for the Treatment Day to proceed. On Treatment Day 2, the average of the FEV1 at 60 minutes and 30 minutes obtained predose must be ≥ 50% and <85% of predicted in order for Treatment Day 2 to proceed.

After the first study drug dose on Treatment Day 1 and on Treatment Day 2, and after each of the following two cumulative doses on each Treatment Day, subjects will undergo spirometry at 5 (+ 2) minutes and at 25 (+/- 2) minutes post-dose. Blood for glucose, potassium and PK sample will be collected at 15 (+/- 5) minutes after the first study drug dose and after each of the following two cumulative doses and vital signs and ECG will be performed at 15 (+/- 5) minutes after the first study drug dose and after each of the following two cumulative doses. Following the last cumulative study drug dose on each Treatment Day, blood for PK sample will be collected at 10, 20, 45, 120, 180, 240, 300, 360, 480, 600 and 720 minutes after the last dose. After the last cumulative dose, spirometry will be performed at 5 (+ 2) minutes and at 25 (+/- 2) minutes. ECG and vital signs will be performed at 15 (+/-5) minutes after the last cumulative dose. After the last cumulative dose, blood will be collected for glucose and potassium at 45 and 120 minutes. Vital signs (BP and HR) will be measured hourly after the last cumulative dose up to 360 minutes and at 480, 600, and 720 minutes after the last dose. The time of each study drug dose will be recorded as the time of the last inhalation of study drug for each individual cumulative dose administered when multiple inhalations are required to administer the dose.

After Treatment Day 2, subjects will be assessed at an End-of-Study (EOS) that will occur 1 to 5 days after the day of the last administration of study drug.

ELIGIBILITY:
Inclusion Criteria:

1. Has provided written informed consent
2. Speaks and understands the English language
3. Males or females 18 to 55 years of age (inclusive) at the Consent Visit
4. Nonsmoker or ex-smoker who has abstained from smoking for at least 1 year prior to the Consent Visit and who has a < 10 pack/year history of lifetime cigarette use
5. Has no history of use of nicotine gum, nicotine patch, e-cigarettes/vaping preparations in the 3 months before the Consent Visit
6. Has a body mass index (BMI) of 18.5 to 40.0 (calculated as kg/m2)
7. Has stable (for at least 6 months) physician-diagnosed asthma with historical documentation of the diagnosis
8. Must be receiving one (1) of the following required inhaled asthma therapies listed below for at least 30 days prior to the Screening Visit: (1) only SABA, which is used for rescue, or (2) low to medium doses of ICS (alone or in combination with SABA and/or LABA), used regularly as maintenance asthma therapy
9. Demonstrates acceptable spirometry performance (i.e., meets American Thoracic Society [ATS]/European Respiratory Society [ERS] acceptability/repeatability criteria
10. Has a pre-bronchodilator FEV1 of ≥50 to <85% of predicted normal value after withholding SABA ≥ 8 hours and (if applicable) LABA for 48 hours
11. Has confirmed FEV1 reversibility to inhaled Ventolin HFA aerosol 180 mcg, defined as a post-Ventolin increase in FEV1 of ≥15 % at or before 30 minutes postdose - NOTE: only 2 reversibility attempts are allowed and, if applicable, a second attempt must occur at least 24 hours after the first attempt and within the 21-day Screening Period
12. Ability to maintain a peak inspiratory flow rate of at least 60 L/min measured by the In-check DIAL device at the medium low resistance setting at the Screening Visit.
13. At the Screening Visit, demonstrates adequate understanding of and ability to successfully inhale from an MDI as determined by the investigator and through demonstrated successful use of the Vitalograph® (Lenexa, KS) aerosol inhalation monitor (AIM™) (training/validation device for MDI) using a placebo MDI canister.

    [Note: potential subjects who cannot demonstrate successful MDI technique using with the AIM device (with placebo canister) after in-clinic training at the Screening Visit will not be eligible for continued participation in the study.]
14. At the Screening Visit, demonstrates adequate understanding of and ability to successfully inhale when using the Halix™ UDDI [Note: a placebo UDDI not containing any drug powder will be supplied for each potential subject to become familiar with the inhaler and practice inhalation technique] [Note: potential subjects who cannot demonstrate successful inhalation technique using the Halix™ UDDI after in-clinic training at the Screening Visit will not be eligible for continued participation in the study].
15. Willing and able to comply with all aspects of the study protocol including avoiding use of certain concomitant medications and attending the required clinic visits (i.e., has no conflicting plans that would prohibit attendance at scheduled study visits including each of the 2 Treatment Day Visits)

    -

Exclusion Criteria:

1. Female subjects of childbearing potential (CBP) who are not using reliable contraception (e.g., abstinence, double barrier method, oral/implantable/transdermal contraception, Depo-Provera, intrauterine device, having one male sexual partner who has undergone vasectomy); a woman is of CBP unless she is premenarchal, is at least 2 years postmenopausal, is without a uterus and/or both ovaries, has had a bilateral tubal ligation, or has undergone the Essure procedure with confirmation of tubal blockage.

   [Note: If a female is identified as less than 2 years postmenopausal, a serum follicle-stimulating hormone (FSH) determination will be performed as a part of screening laboratory assessments. If an FSH result of < 40 mIU/mL is obtained, the female will be determined to be of CBP and her unwillingness to use reliable contraception as defined above will be exclusionary for the study.]
2. A woman who is pregnant (has a positive serum pregnancy test at Screening Visit), is lactating, or is likely/planning to become pregnant during the study
3. Vital signs at the Screening Visit (after at least 2 minutes seated at rest) showing SBP either < 80 mmHg or >150 mmHg; DBP > 90 mmHg; or HR either < 40 bpm or > 100 bpm (vital signs outside these criteria may be repeated once after an additional seated rest period of at least 2 minutes- if vital signs exclusion criteria are not met after the repeat measurements of SBP, DBP, or HR, screening may continue)
4. Chronic obstructive pulmonary disease or other significant lung disease (e.g. chronic bronchitis, emphysema, bronchiectasis with a need for treatment, cystic fibrosis, or bronchopulmonary dysplasia)
5. Oral corticosteroid use at any dose within the 6 weeks prior to the Screening Visit
6. Receipt of any marketed (e.g. omalizumab, mepolizumab, reslizumab) or investigational biologic within 3 months of the date of the Screening Visit or within 5 half-lives of the drug, whichever is longer
7. Currently a smoker, or a former smoker with > 10 pack-year history, or a former smoker who stopped smoking <1 year before the Screening Visit
8. A history of life-threatening asthma defined as any history of significant asthma episodes(s) requiring intubation associated with hypercapnia, respiratory arrest, hypoxic seizures, or asthma-related syncopal episode(s)
9. Emergency room visit or hospitalization for any acute respiratory condition in the 3 months prior to the Screening Visit
10. Current history of uncontrolled hypertension or uncontrolled diabetes, in the opinion of the Investigator (NOTE: controlled hypertension and/or controlled diabetes are not exclusionary)
11. Presence of cancer not in remission for at least 5 years prior to the Screening Visit (excludes non-melanomatous skin cancer)
12. Hospitalized for psychiatric disorder in the previous 12 months or has a history of attempted suicide within 5 years prior to the Screening Visit
13. Unable to abstain from protocol-defined prohibited medications during the study
14. Clinical laboratory tests (after ≥4 hours fasting) at the Screening Visit that show results outside the normal ranges for the following clinical laboratory tests that, in the Investigator's opinion, are judged to be clinically significant:

    * hemoglobin
    * hematocrit
    * total white blood cell count (WBC)
    * platelet count
    * serum glucose
    * serum potassium
    * ALT
    * AST
    * alkaline phosphatase
    * serum creatinine
15. Clinical laboratory tests at the Screening Visit that show any of the following:

    * positive serum hCG (female subjects only)
    * positive urine drug screen (exception is evidence of authorized prescribed medications)
    * positive urine cotinine test
16. Presence of any uncontrolled (in the Investigator's medical opinion) systemic disease, including, but not limited to renal, hepatic, hematologic, gastrointestinal, endocrine, pulmonary, cardiac, neurologic, or psychiatric disease
17. Electrocardiogram obtained at Screening Visit that shows (in the Investigator's medical opinion) medically significant abnormalities (e.g., left bundle branch block, frequent premature ventricular contractions, chronic atrial fibrillation, or QTcB interval prolongation > 450 msec for males and > 470 msec for females)
18. Presence of current drug or alcohol abuse, in the Investigator's opinion, making it unlikely that the requirements of the subject's participation in the protocol will be met
19. History of allergic reaction (known hypersensitivity) to albuterol sulfate and/or lactose, in any formulation
20. History of intolerance to aerosolized β2-adrenergic agonists
21. Receipt of a drug or biologic in an investigational research study within the 30 days prior to the Screening Visit
22. An elective surgical or medical procedure currently is planned or scheduled to be performed during the study (this excludes routine immunotherapy/desensitization procedures that are being performed on a regular schedule and have been unchanged for at least 3 months prior to the Screening Visit)
23. Presence of a clinically diagnosed upper respiratory tract infection within the 7 days prior to the Screening Visit

    -

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2018-06-30 (Actual); Primary Completion 2018-08-31 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
Analyses of baseline-adjusted FEV1 (liters) at 25 (+/- 2) minutes after each initial and cumulative dose of albuterol | At each of the treatment visits, FEV1 will be measured prior to initial drug administration and at 25 minutes after each cumulative and hourly up to 6 hours after last dose
  Change from treatment day baseline in forced expiratory volume in one second (FEV1) (liters) will be assessed at 25 minutes after each cumulative dose of albuterol and serially up to 360 minutes after the last dose

SECONDARY OUTCOMES:
Analyses of baseline-adjusted FEV1 at 5 (+2) minutes after each initial and cumulative dose of albuterol | At each of the two treatment visits, FEV1 (forced expiratory volume in one second) will be measured prior to initial drug administration and at 5 minutes after each cumulative dose adminstered at 30 minute intervals and up to 6 hours after the last dose
  Change from treatment day baseline in forced expiratory volume in one second (FEV1) will be assessed at 5 minutes after each cumulative dose of albuterol and serially up to 360 minutes after the last dose of albuterol
Baseline-adjusted FEV1 AUC0-6 (liter-hour) after the last cumulative dose of albuterol | At each of the treatment visits, FEV1 will be measured hourly from after the last dose of albuterol until 6 hours post-dose
  Area under the efficacy curve (AUC) for the period of 0 to 6 hours after the last dose of albuterol
Comparison of the FEV1 at the lowest dose of albuterol and the highest cumulative dose of albuterol for each drug/device | At each of the treatment visits, FEV1 (liters) will be measured prior to the first dose of albuterol and at 5 and 25 minutes after each dose of albuterol
  Change from treatment day baseline in FEV1 will be assessed at 5 and 25 minutes after the first dose of albuterol and at 5 and 25 minutes after the last dose of albuterol to assess the dose-response for each drug/device evaluated
Systolic and diastolic blood pressure (mmHg) before and after each dose of albuterol | Serial measurements of systolic and diastolic blood pressure in mmHg will be taken at baseline on each treatment day, at 15 minutes after each dose of albuterol, and at each hour post-dose for 6 hours after the last dose of albuterol
  Change from treatment day baseline in sytolic and diastolic blood pressure (mmHg) will be evaluated by the maximum change in mmHg (systolic and diastolic) and minimum change in mmHg (systolic and diastolic) from baseline blood pressures, and the
  weighted mean change (in mmHg) from baseline in systolic and diastolic blood pressure
Heart rate (beats per minute) before and after each dose of albuterol | Serial measurements of heart rate (beats per minute) will be taken at baseline on each treatment day, at 15 minutes after each dose of albuterol, and at each hour for 6 hours after the last dose of albuterol
  Change from treatment day baseline in heart rate (beats per minute) will be evaluated by the maximum change in beats per minute and minimum change in beats per minuet from baseline heart rate, and the
  weighted mean change in beats per minute from baseline in heart rate
Serum potassium and glucose before and after each dose of albuterol | Serial measurments of serum potassium (mg/dL) and glucose (mg/dL) will be obtained pre-dose and at at 10-20 minutes after each dose of albuterol up to and including 2 hours after the last dose of albuterol
  Change from baseline serum potassium (mg/dL) and glucose (mg/dL) will be evaluated by the description of changes in mg/dL from baseline values
Electrocardiographic QTc interval (milliseconds) before and after inhalation of initial and cumulative doses of albuterol | Serial ECGs (electrocardiograms) will be obtained before the first albuterol dose on each treatment day, at 15 minutes after each albuterol dose, and at hourly intervals up to 6 hours after the last albuterol dose
  Change from treatment day baseline ECG (electrocardiogram) will assess the maximum and mean change from baseline of the corrected QT interval in milliseconds (QT measures the time between the start of the Q wave and the end of the T wave in the heart's electrical cycle) following each of the doses of albuterol
Assessment of adverse events following administration of albuterol | At each of the treatment visits, spontaneously reported adverse events will be assessed continually during the time subject is in clinic up to approximately 15 hours after first dose of albuterol
  Incidence, type, and severity of adverse events reported after each of two cumulative dose regimens of albuterol

OTHER OUTCOMES:
Peak plasma concentrations of albuterol after oral inhalation on each of 2 treatment days | PK samples will be collected at approximately 15 minutes after each dose of albuterol and at hourly intervals up to 720 minutes after the last dose of albuterol on each treatment day
  Sample for plasma albuterol concentration will be obtained before the first dose of albuterol on each treatment day and after each of the cumulative doses of albuterol
Area under the plasma concentration versus time (AUC0-t) for albuterol after inhalation of cumulative doses of albuterol at 30 min intervals | PK samples will be collected at approximately 15 minutes after each dose of albuterol and at hourly intervals up to 720 minutes after the last dose of albuterol
  Pre-dose and post dose measurement of albuterol in plasma will be assessed after each dose of albuterol on each treatment day

CONTACTS AND LOCATIONS:
Locations (1):
- North Carolina Clinical Research, Raleigh, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No